CLINICAL TRIAL: NCT00482846
Title: Phase I Dose Escalation Trial of High Dose Melphalan Conditioning Regimen With Palifermin for Cytoprotection Followed by Autologous Peripheral Blood Stem Cell Transplantation for Multiple Myeloma
Brief Title: Melphalan and Palifermin in Treating Patients Undergoing An Autologous Peripheral Stem Cell Transplant for Stage II or III Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Muneer Abidi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000547155; P30CA022453 (NIH); WSU-2006-119; NCT01654744 (obsolete NCT alias)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Mucositis; Multiple Myeloma
Keywords: mucositis; drug/agent toxicity by tissue/organ; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Mucositis; Multiple Myeloma; Drug-Related Side Effects and Adverse Reactions | interventions — Fibroblast Growth Factor 7; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palifermin & Melphalen (Experimental): Palifermin 60 mcg/kg/d of the actual body weight unless actual body weight is >40% of the Ideal body weight (IBW), then adjusted body weight (AdBW) will be used for dose calculations - administered on Day - 5,-4, - 3 and then repeated on Day +1, +2 and +3
  Dose of Melphalan + Palifermin (Normal Renal Function): All given on Day -2:
  Dose Level 1- 200 mg/m2 I.V; Dose Level 2- 220 mg/m2 I.V; Dose Level 3- 240 mg/m2 I.V; Dose Level 4- 260 mg/m2 I.V; Dose Level 5- 280 mg/m2 I.V;
  Dose of Melphalan + Palifermin (Renal Dysfunction CrCl. <60)adm. via I.V.:
  Dose Level 1- 140 mg/m2; Dose Level 2- 160 mg/m2; Dose Level 3- 180 mg/m2; Dose Level 4- 200 mg/m2; Dose Level 5- 220 mg/m2;
  Interventions: Biological: Palifermin; Drug: melphalan; Other: questionnaire administration; Procedure: autologous peripheral blood stem cell transplantation; Other: quality-of-life assessment

INTERVENTIONS:
Biological: Palifermin — Palifermin 60 mcg/kg/d of the actual body weight unless actual body weight is >40% of the Ideal body weight (IBW), then adjusted body weight (AdBW) will be used for dose calculations - administered on Day - 5,-4, - 3 and then repeated on Day +1, +2 and +3
  Other Names: Kepivance
Drug: melphalan — Dose of Melphalan + Palifermin (Normal Renal Function): All given on Day -2:
  Dose Level 1- 200 mg/m2 I.V; Dose Level 2- 220 mg/m2 I.V; Dose Level 3- 240 mg/m2 I.V; Dose Level 4- 260 mg/m2 I.V; Dose Level 5- 280 mg/m2 I.V;
  Dose of Melphalan + Palifermin (Renal Dysfunction CrCl. <60)adm. via I.V.:
  Dose Level 1- 140 mg/m2; Dose Level 2- 160 mg/m2; Dose Level 3- 180 mg/m2; Dose Level 4- 200 mg/m2; Dose Level 5- 220 mg/m2;
  Other Names: Alkeran
Other: questionnaire administration — Day -5 to Day +28
Procedure: autologous peripheral blood stem cell transplantation — Day 0
Other: quality-of-life assessment — Day -5 to Day +28

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Keratinocyte growth factors, such as palifermin, may help prevent symptoms of mucositis, or mouth sores, in patients receiving melphalan before a peripheral stem cell transplant for multiple myeloma.

PURPOSE: This phase I trial is studying the side effects and best dose of melphalan when given together with palifermin in treating patients undergoing an autologous peripheral stem cell transplant for stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of high-dose melphalan when administered with palifermin in patients undergoing autologous peripheral blood stem cell transplantation for stage II or III multiple myeloma.

Secondary

* Assess overall response (complete and partial response and stable disease) in these patients at 28 and 100 days post-transplantation.
* Assess the efficacy of palifermin as a cytoprotective agent in reducing incidence and duration of mucositis in patients treated with this regimen.
* Assess patient-reported outcomes and impact of palifermin on quality of life of these patients.
* Assess the qualitative and quantitative toxicities of this regimen in these patients.

OUTLINE: This is a dose-escalation study of melphalan. Patients are stratified according to creatinine clearance (normal vs < 60 mL/min).

Patients receive high-dose melphalan IV on day -2 and palifermin IV on days -5 to -3 and 1-3. Patients undergo autologous peripheral blood stem cell transplantation on day 0.

In each stratum, cohorts of 3-6 patients receive escalating doses of melphalan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients complete questionnaires about overall health, mouth and throat soreness (MTS), and activity limitations due to MTS once daily on days -5 to 28.

After completion of study treatment, patients are followed at days 28 and 100 and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Stage II or III disease
* Must have undergone successful stem cell mobilization (≥ 2.0 x 10^6 CD34+ cells/kg)
* No oral lesions from any other etiology
* No unhealed mucositis from induction treatment

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Amylase and lipase normal
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Creatinine normal (stratum 1 only)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV positivity
* No history of allergic reaction attributed to melphalan
* No uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* No hepatitis B or C positivity
* No prior or concurrent pancreatitis
* No known sensitivity to any of the study drugs, including E. coli-derived products

PRIOR CONCURRENT THERAPY:

* Prior bone marrow or stem cell transplantation allowed
* No prior palifermin
* More than 30 days since prior investigational agents
* No concurrent dialysis
* No concurrent amifostine
* No concurrent prophylactic oral cryotherapy during melphalan administration
* No concurrent mouthwash solutions containing any of the following:

  * Chlorhexidine
  * Hydrogen peroxide
  * Diphenhydramine hydrochloride
* No concurrent recombinant interleukin-11 or sargramostim (GM-CSF)
* No concurrent sucralfate in suspension form

  * Sucralfate tablets allowed
* No concurrent povidone-iodine rinses
* No concurrent glutamine as a prophylactic agent for mucositis
* No other concurrent investigational agents
* No concurrent antithymocyte globulin suppression or alemtuzumab
* No concurrent rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-06; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of melphalan when treated with palifermin to prevent mucositis | Days -5, -4, -3, 2, +1, +2 and +3

SECONDARY OUTCOMES:
Dose-limiting toxicity | Days -5, -4, -3, 2, +1, +2 and +3
Evaluate the efficacy of Palifermin as a cytoprotective agent in reducing incidence and duration of Grade 3 and 4 mucositis due to high dose Melphlan | Day -5 to Day +28
Overall response | At Day 28 and Day100 after autologous transplant when treated with combination of palifermin and Melphalan
Reduction in incidence and duration of mucositis | Days -5 to Day +28

CONTACTS AND LOCATIONS:
Overall Officials: Muneer H. Abidi, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States